CLINICAL TRIAL: NCT01687062
Title: Iron Absorption From Tef-injera in Women of Reproductive Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EK2012N31
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Iron Deficiency
Keywords: NaFeEDTA; phytate; injera; iron absorption
MeSH Terms: conditions — Iron Deficiencies | interventions — Fe(III)-EDTA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- FeSO4 + high phytate (Active Comparator): injera test meal 1 labeled with a 4 mg staple iron isotope tag
  Interventions: Other: FeSO4
- FeSO4 + medium phytate (Experimental): injera test meal 2 labeled with a 4 mg staple iron isotope tag
  Interventions: Other: FeSO4; Other: reduction of phytate
- FeSO4 + low phytate (Experimental): injera test meal 3 labeled with a 4 mg staple iron isotope tag
  Interventions: Other: FeSO4; Other: reduction of phytate
- FeSO4 + NaFeEDTA (1:1) + high phytate (Experimental): injera test meal 4 labeled with a 4 mg staple iron isotope tag
  Interventions: Other: FeSO4; Other: NaFeEDTA
- FeSO4 + NaFeEDTA (1:3) + high phytate (Experimental): injera test meal 5 labeled with a 4 mg staple iron isotope tag
  Interventions: Other: FeSO4; Other: NaFeEDTA

INTERVENTIONS:
Other: FeSO4
Other: reduction of phytate
  Arms: FeSO4 + low phytate; FeSO4 + medium phytate
Other: NaFeEDTA
  Arms: FeSO4 + NaFeEDTA (1:1) + high phytate; FeSO4 + NaFeEDTA (1:3) + high phytate

SUMMARY:
Anemia is one of the most common health problems all over the world with around half of preschool-aged children (<5 years) and one third of women affected. Nutritional iron deficiency is a major reason for anemia in infants, young children and women of reproductive age who have especially high iron requirements that are difficult to meet in regions where the major diet is based on plant foods. So in Ethiopia, where injera is the major staple food. Despite high levels of iron in tef, the most favored cereal for injera, the iron bioavailability is assumed to be very low due to the high levels of phytic acid found in tef.

The aim of this study is to determine the iron bioavailability in women from injera prepared in a traditional way and investigate the potential of methods to improve the bioavaiability. Therefore, a 50/50 and a 25/75 blend of FeSO4 and NaFeEDTA for iron fortification will be evaluated. Further the potential positive impact of phytic acid reduction on the iron bioavailability will be investigated. The phytic acid reduction will be achieved in two different ways, by addition of whole grain wheat as source of phytase and addition of a commercially available microbial phytase. The studies will be conducted in healthy women using stable isotope techniques.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age females 18-40 years
* Maximum body weight 65 kg
* Normal body mass index (18.5-25 kg/m2)
* No intake of mineral/vitamin supplements 2 weeks before and during the study
* No metabolic or gastrointestinal disorders or chronic diseases
* Not pregnant or lactating
* No regular intake of medication (except oral contraceptives)
* No blood donation or significant blood loss (accident, surgery) over the past 4 months
* Not currently participating in another clinical trial or having participated in another clinical trial during the last 3 months prior to the beginning of this study
* No former participation in a study involving administration of iron stable isotopes
* No eating disorders or food allergy
* Subject who can be expected and are willing to comply with study protocol
* Having received oral and written information about the aims and procedures of the study
* Having provided oral and written informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Iron absorption | 17 days
  Test meals with isotopic iron labels will be administrated on day 1-3. Whole blood samples will be collected on day 17 (14 after the last test meal) to analyze the iron isotope ratios.

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Switzerland